CLINICAL TRIAL: NCT06356688
Title: A Clinical Study on the Efficacy and Safety of Paclitaxel Polymeric Micelles for Injection and Cisplatin Combined With Cadonilimab as a Neoadjuvant Therapy for Locally Advanced Esophageal Squamous Cell Carcinoma: A Single-Arm, Single-Center, Prospective Clinical Trial (POINTS Trial)
Brief Title: A Clinical Study on the Efficacy and Safety of Paclitaxel Polymeric Micelles and Cisplatin Combined With Cadonilimab as a Neoadjuvant Therapy for Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Jing (Other)
Responsible Party: Sponsor-Investigator, Sun Jing, chief physician、professor, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13914704178
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapy
Keywords: cadonilimab; neoadjuvant therapy; esophageal squamous cell carcinoma; Paclitaxel Polymeric Micelles for Injection
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Paclitaxel Polymeric Micelles for Injection and Cisplatin combined with Cadonilimab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel Polymeric Micelles for Injection and Cisplatin Combined with Cadonilimab (Experimental)
  Interventions: Drug: Paclitaxel Polymeric Micelles for Injection and Cisplatin combined with Cadonilimab

INTERVENTIONS:
Drug: Paclitaxel Polymeric Micelles for Injection and Cisplatin combined with Cadonilimab — Paclitaxel Polymeric Micelles for Injection:Cycle 1: 230mg/m2, IV ≥3 hours; Cycles 2-4: If the patient has a neutrophil nadir ≥1.0 x 109/L along with a platelet nadir ≥80 x 109/L after Cycle 1 dosing and has not experienced grade II-IV non-hematologic toxicity, then give 260mg/m2, IV ≥3 hours, d1, q3w; Cisplatin: 25mg/m2/d x d1-3, IV drip, q3w; Cadonilimab: 10mg/kg, IV drip, d3, q3w;

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of neoadjuvant treatment of locally advanced esophageal squamous carcinoma with a PD-1/CTLA-4 bispecific antibody (Cadonilimab) in combination with platinum-containing chemotherapy (Paclitaxel Polymeric Micelles for Injection combined with Cisplatin). Includes pathologic complete remission rates (pCR rates) after 2-4 cycles of Cadonilimab combination chemotherapy. The objective remission rate (ORR), major pathologic remission rate (MPR), R0 resection rate and 2-year overall survival (OS) and progression-free survival (OS) rates, and safety of neoadjuvant treatment of locally advanced esophageal squamous carcinoma with Cadonilimab combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, ≤75 years, gender is not limited;
2. Squamous esophageal cancer of thoracic segment confirmed by pathology;
3. Locally advanced patients with no distant metastasis by imaging, resectable or potentially resectable after discussion among oncology, esophageal surgery, and imaging, and clinical stage cT2-4aN+ or cT3-4aN0, M0, stage II, III, or IVA (AJCC 8th edition cTNM staging);
4. ECOG PS score of 0-1;
5. No previous antitumor treatment such as radiotherapy, chemotherapy and immunotherapy;
6. Expected survival > 6 months;
7. Adequate baseline organ function: (i) WBC ≥3×10^9/L, ANC ≥1.5×10^9/L, PLT ≥100×10^9/L, Hb ≥9g/dL; (ii) Liver function: TBIL ≤2ULN, AST ≤2.5ULN, ALT ≤2.5ULN; (iii) Renal function: cCr>40 ml/min, Cr≤1.5 ULN; (iv) Cardiac function: no cardiac disease or coronary artery disease. Cardiac function: no heart disease or coronary heart disease, patients with cardiac function grade 1-2;
8. Hypertensive patients applying antihypertensive drugs to control blood pressure within the normal range;
9. Diabetic patients with fasting blood glucose controlled at ≤8mmol/L by hypoglycemic drug treatment;
10. No other serious diseases (such as autoimmune diseases, immunodeficiency, organ transplantation, or other diseases that require continuous hormone therapy) that conflict with this protocol;
11. No history of other malignant tumors;
12. The patient agrees to participate in this clinical study and signs the Informed Consent Form.

Exclusion Criteria:

1. Patients who have previously received anti-tumor therapy (including chemotherapy, radiotherapy, surgery or immunotherapy, etc.);
2. Combination of other incurable malignant tumors (except cured non-malignant skin tumors, cervical cancer in situ, and prostate cancer);
3. Patient has or anticipates a significant risk of esophageal perforation, fistula, and hemorrhage;
4. Active autoimmune or immunodeficiency disease, use of immunosuppressants prior to enrollment, and use of immunosuppressant dosage ≥10 mg/day of oral prednisone for more than 2 weeks;
5. Clinically significant cardiovascular disease including, but not limited to, severe acute myocardial infarction, unstable or severe angina pectoris, coronary artery bypass grafting surgery, congestive heart failure, ventricular arrhythmia requiring medical intervention, left ventricular ejection fraction <50%, or other anticipated inability to tolerate chemoradiotherapy in the 6 months prior to enrollment;
6. Severe allergies;
7. Pregnant or lactating women;
8. Severe mental disorders;
9. Presence of CTC grade ≥3 peripheral nerve disease;
10. Abnormal coagulation function (PT > 16s, APTT > 53s, TT > 21s, Fib < 1.5g/L), bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
11. Presence of severe pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, severe impairment of lung function, or active tuberculosis within 1 year;
12. Presence of active hepatitis B or C;
13. Any other condition that the investigator evaluates to be ineligible for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rates | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  evaluate pathological complete response rate of primary tumor and locally metastatic lymph nodes after 2-4 cycles of neoadjuvant therapy.

SECONDARY OUTCOMES:
Objective Rate of Effectiveness (ORR) | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  the proportion of patients who achieve PR or CR
R0 Removal Rate | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Rate of microscopically margin-negative resection
2-year overall survival rate | 2 years
  2-year overall survival rate
2-year disease free survival rate | 2 years
  2-year disease free survival rate
major pathological response (MPR) | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No